CLINICAL TRIAL: NCT04198441
Title: A Randomized, Multicenter, Open Label Study Comparing the Omeza® Products Bundle to Standard of Care for Chronic Venous Leg Ulcers and Chronic Diabetic Foot Ulcers
Brief Title: The Omeza Protocol for Chronic Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Number: 100
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Venous Leg Ulcer; Diabetic Foot Ulcer
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Omeza Value-based Bundle Test (Active Comparator): The Omeza value-based bundle consists of lidocaine lavage, flowable collagen matrix and skin protectant products.
  Interventions: Device: Wound dressing
- Standard Wound Care Control (Active Comparator): Standard wound care control is saline wound wash and wet to dry dressing.
  Interventions: Device: Wound dressing

INTERVENTIONS:
Device: Wound dressing — Clean wound, fill wound, dress wound

SUMMARY:
This study will compare the Omeza® Products Bundle to standard of care (SOC) for in subjects with chronic venous leg ulcers and subjects with diabetic foot ulcers.

DETAILED DESCRIPTION:
This is a randomized, multi-center, open-label study comparing the Omeza® Products Bundle versus standard of care treatments for 2 different types of chronic ulcers (venous leg ulcers and diabetic foot ulcers). The treatment period will be 12 weeks, with subjects coming into the study site weekly for evaluations, photography and formal measurements of the target wound, and dressing changes. There will be a total of 13 study site visits. The Screening Visit (Day 0) will occur 1 week prior to randomization and will include routine labs and vascular assessment to determine inclusion/exclusion of the potential subject from the study; followed by weekly treatment visits (Week 1 through Week 11); randomization will occur at Treatment Visit Week 1; the Treatment Visit Week 12/End of Study Visit will include end of study labs. Target wounds will be photographed and measured, and vascular assessment will be done at each of the 13 visits.

If the wound closes before Week 12, the subject will continue to come in for all the remaining study visits until study completion. If the wound does not close by Week 12, the subject will be immediately exited from the study and no further follow-up will occur as part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 21-80 years of age
2. Participated in the informed consent process and signed study specific informed consent document
3. Willing and able to comply with study procedures, including study visits and study dressing regimens
4. Confirmation of venous disease by non-invasive venous studies with either Doppler- confirmed venous reflux or having ≥ 2 clinical characteristics of venous insufficiency (varicose veins, lipodermatosclersosis, venous dermatitis, atrophie blanche, edema). Biopsy done to exclude other skin conditions e.g. cancer on ulcers ≥ 6 months
5. HbA1c of ≤ 10%
6. Have a venous ulcer between the knee and ankle, at or above the malleolus
7. For VLU's: Target wound size ≥ 4 cm2 to ≤ 150 cm2 in area without exposed tendon, muscle or bone For DFU's: Target wound size ≥ 0.25 cm2 to ≤ 150 cm2 post debridement at Screening Visit and Treatment Visit Week 1/Randomization
8. Target wound duration of at least 3 months and less than or equal to 12 months as of the date the subject signs consent for study
9. Containing yellow/white slough with or without fibrous/scar tissue and/or non- viable tissue
10. Be willing and able (or have family member/friend willing and able) to apply required dressing changes as well as the ability of the subject to tolerate limb compression bandage
11. Ankle-Branchial Index (ABI) less than 0.80 or greater than 1.3

Exclusion Criteria:

1. Subjects with a BMI ≥ 65
2. Subject is medically unable to consent (due to head trauma, coma, etc.) or cognitively impaired (due to being mentally challenged, having Alzheimer

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 13 weeks
  Percent wound closure from baseline
Wound Closure Rate | 13 weeks
  Rate of wound closure measured weekly
Time to Maximum Wound Closure | 1-13 weeks
  Number of weeks to achieve complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Applewhite, MD,CWSP,FUHM, Principal Investigator — Baylor University Medical Center's Comprehensive Wound Center; David Swain, DPM,CWSP, Principal Investigator — First Coast Cardiovascular Institute; Robert B McLafferty, MD,MBA,FACS, Principal Investigator — Oregon Health and Science University; Jacob Reinkraut, DPM,FACFAS, Principal Investigator — Saint Michael's Medical Center
Locations (4):
- United States (4):
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Saint Michael's Medical Center, Newark, New Jersey
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Baylor Scott & White Comprehensive Wound Care Center, Dallas, Texas